CLINICAL TRIAL: NCT03253276
Title: Effect of Obeticholic Acid (INT-747, Intercept) on the Hepatobiliary Transport of Bile Acids in Patients With PBC Examined by 11C-cholyl-sarcosine PET/CT
Brief Title: Effect of Obeticholic Acid on Transport of Bile Acids in PBC Examined by 11C-cholyl-sarcosine PET/CT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: OCAPBC
Record Dates: First submitted 2017-05-28; First posted 2017-08-17 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Bile Acid Transporter
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — obeticholic acid

STUDY DESIGN:
Intervention Model Description: Double blind placebo-controlled crossover
Who Masked: Participant, Investigator
Masking Description: Codes (OCA or placebo) will be opened after final examination of final patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obeticholic Acid (Active Comparator): Patients with primary biliary cirrhosis are treated 3 months with OCA (active drug) or placebo in a double-blind cross-over study design.
  Interventions: Drug: Obeticholic acid
- placebos (Placebo Comparator): Patients with primary biliary cirrhosis are treated 3 months with OCA (active drug) or placebo in a double-blind cross-over study design.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Obeticholic acid — Placebo-controlled
  Other Names: placebo
  Arms: Obeticholic Acid
Drug: Placebos
  Other Names: Obeticholic acid
  Arms: placebos

SUMMARY:
This is an investigator-initiated, double-blind crossover study on the mechanism of OCA treatment of patients with PBC.

Hypothesis and significance

The investigators will test the hypothesis that OCA administration to patients with PBC increases hepatobiliary secretion of cholylsarcosine assessed by PET/CT using 11C-labeled cholylsarcosine (11C-CSar) as tracer.

The results of this research project will elucidate the mechanism of the effect of using OCA therapeutically in patients with PBC.

DETAILED DESCRIPTION:
Background

Primary biliary cholangitis (PBC) is a chronic autoimmune liver disease characterized by cholestasis and cirrhosis. Pathogenesis comprises impaired hepatobiliary secretion of bile acids to the bile. As a result bile flow reduces and diminished content of bile acids in the intestines leads to impaired absorption of lipids and lipid-soluble vitamins, diarrhea, general pruritus, and fatigue.

Bile acids are transported from blood to hepatocytes by the transporter proteins Na+-taurocholate co-transporting polypeptide (NTCP) and Organic anion-transporting polypeptide (OATP) and secreted from hepatocyte to bile canaliculi by the Bile salt export pump (BSEP) and Multidrug resistance protein type 3 (MDR3). Dysfunction of BSEP most probably plays a key pathogenic role in PBC.

Ursodeoxycholic acid (UDCA) is a dihydroxylated bile acid and the only approved drug for treatment of PBC today. In most cases UDCA can delay or prevent disease progression. However, a subgroup of patients does not respond adequately to UDCA and for these patients new therapies are needed.

BSEP is induced by the nuclear bile acid receptor (BAR), also known as farnesoid X receptor (FXR). Obeticholic Acid (INT-747, Intercept) (OCA) is a FXR agonist and induces BSEP.

OCA administration therefore may increase the hepatobiliary secretion of bile acids, being the mechanism behind beneficial therapeutic effects in PBC.

Cholylsarcosine is a synthetic conjugated bile acid (sarcosine = methyl-glycine) that is non-toxic, not metabolized in the gut or liver, and transported by BSEP. The trans-hepatic transport of bile acids can be assessed in humans by PET/CT of the liver using 11C-labeled cholylsarcosine (11C-CSar) as tracer. 11C-CSar is handled by the liver as a natural bile acid in pig studies (1). Studies in humans (2) show that

* 11C-CSar is taken up avidly by the liver and flow-determined
* 11C-CSar secretion from hepatocytes to bile is reduced during cholestasis, and
* 11C-CSar back flux from hepatocytes to blood during cholestasis

Patients

8 patients with PBC

* who are not responding adequately to treatment with UDCA, defined as ALP > 2 times upper normal level during a time period of 6 months
* Patients are recruited from Aarhus University Hospital, Department of Hepatology and Gastroenterology.

Paired study design

* 11C-CSar PET/CT before and after 3 months treatment with OCA or placebo.

Methods

PET/CT: Initial low-dose CT for anatomical definition of the PET findings and for attenuation correction of PET data. Dynamic 60-min PET recording of the tissue radioactivity concentration over time following iv bolus injection of 100 MBq 11C-CSar and iv infusion of 100 MBq 11C-CSar. During the PET study, ICG is given as a constant iv infusion for measurements of hepatic blood flow, used in the kinetic analysis, and blood samples are collected from catheters in a radial artery and a liver vein (blood 11C-CSar concentrations for kinetic calculations, ICG, and blood gasses for monitoring purposes).

Liver tests at the time points of the PET/CT study: Plasma ALT, ALP, GGT, bilirubin, bile salts, IRN, platelets, hemoglobin, mitochondrial antibodies; ICG clearance.

Raw data comprise time-courses of the 11C-CSar concentrations in liver tissue and common hepatic bile duct (PET recordings) and blood concentrations of 11C-CSar in arterial and liver vein blood (blood samples); hepatic blood flow, hepatic venous pressure gradient (HVPG), splanchnic oxygen uptake.

11C-CSar data comprise clearances of 11C-CSar from blood-to-hepatocytes and from hepatocytes-to-bile canaliculi, vascular extraction fractions, biliary secretion fraction, transit times, etc.

ELIGIBILITY:
Inclusion Criteria:

* patients with PBC
* who are not responding adequately to treatment with UDCA, defined as ALP > 2 times upper normal level during a time period of 6 months

Exclusion Criteria:

* Itching that requires medical treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Effect of OCA on bile flow | Measured after 3 months of treatment with Obeticholic Acid or placebo
  Bile flow measured by PET

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Keiding, prof, Principal Investigator — University of Aarhus
Locations (1):
- Susanne Keiding, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Orntoft NW, Munk OL, Frisch K, Ott P, Keiding S, Sorensen M. Hepatobiliary transport kinetics of the conjugated bile acid tracer 11C-CSar quantified in healthy humans and patients by positron emission tomography. J Hepatol. 2017 Aug;67(2):321-327. doi: 10.1016/j.jhep.2017.02.023. Epub 2017 Feb 27. PMID 28249726
- [Result] Sorensen M, Munk OL, Orntoft NW, Frisch K, Andersen KJ, Mortensen FV, Alstrup AK, Ott P, Hofmann AF, Keiding S. Hepatobiliary Secretion Kinetics of Conjugated Bile Acids Measured in Pigs by 11C-Cholylsarcosine PET. J Nucl Med. 2016 Jun;57(6):961-6. doi: 10.2967/jnumed.115.171579. Epub 2016 Mar 10. PMID 26966160
- [Result] Frisch K, Jakobsen S, Sorensen M, Munk OL, Alstrup AK, Ott P, Hofmann AF, Keiding S. [N-methyl-11C]cholylsarcosine, a novel bile acid tracer for PET/CT of hepatic excretory function: radiosynthesis and proof-of-concept studies in pigs. J Nucl Med. 2012 May;53(5):772-8. doi: 10.2967/jnumed.111.098731. Epub 2012 Mar 27. PMID 22454486
- [Derived] Kjaergaard K, Frisch K, Sorensen M, Munk OL, Hofmann AF, Horsager J, Schacht AC, Erickson M, Shapiro D, Keiding S. Obeticholic acid improves hepatic bile acid excretion in patients with primary biliary cholangitis. J Hepatol. 2021 Jan;74(1):58-65. doi: 10.1016/j.jhep.2020.07.028. Epub 2020 Jul 25. PMID 32717289